CLINICAL TRIAL: NCT03445507
Title: Effectiveness of a Chat Bot for Smoking Cessation: a Pragmatic Trial in Primary Care.
Acronym: Dej@lo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Eduardo Olano, Phd in Medicine. Family and Community Medicine Specialist, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17/01942
Record Dates: First submitted 2018-02-06; First posted 2018-02-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco; cessation; medical apps for smartphones
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: N = 460 smokers (230 in each arm), who will be recruited before randomization. Interventions: Intervention group: Use of an evidence-based chat bot for smoking cessation. Control group: Usual care (Madrid Health System Portfolio).
Masking Description: Intervention can´t be masked. We will objectify primary outcome by biochemistry validation, and statistician conducting the analysis will not know to which study arm a given patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of an evidence-based chat bot for smoking cessation
  Interventions: Other: Chat bot
- Control (Active Comparator): Usual care (Madrid Health System Portfolio).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Chat bot — Patients in intervention arm will use an evidence-based chat bot as an aid for smoking cessation
  Other Names: Intervention arm
  Arms: Intervention
Other: Usual care — Usual care given by their usual general practitioners and nurses of primary care health centres, as defined in Public Health System Portfolio.
  Other Names: Active comparator arm
  Arms: Control

SUMMARY:
This study aims to evaluate the effectiveness of an intervention to help people to quit smoking throughout an chat bot compared with usual assistance to increase long-term rates of nicotine abstinence in smoking outpatients with biochemical validation at 6 months.

Half of participants(control group) will receive usual care by their usual general practitioners and nurses, and the other half (intervention group) will use an evidence-based chat bot specifically designed to help people quit smoking.

DETAILED DESCRIPTION:
An array of interventions have been shown to be both cost-effective and efficacious in helping patients quit smoking and so are included in usual care given by general practitioners and nurses. However, in the primary care setting, this sort of interventions are less common than they should be, due to many circunstances, and solutions must be found due to the huge dimensions of tobacco use challenge.

On the other hand,new kinds of information tecnology give a chance to intervene with less costs and more specific tools. Actually, there are a lot of mobile apps and other devices designed to help people to improve their health in many ways, but without scientific evidence of their effects.

This is a pragmatic, randomised, controled and multicentric clinical trial that tries to evaluate in general population the effectiveness of a chat bot that incorporates evidence based interventions and interacts by a text application instaled in patients mobile phone (intervention group).

Investigators have decided to compare with usual care delivered by the usual general practisioners and nurses of Spanish Public Health Centres, because this interventions have shown their effectiveness (control group).

Efficiency and impact on quality of life will also be compared on both groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* Smoked more than one cigarette per day last month.
* Accepts help to quit smoking next month.
* Owns a mobile phone with the ability to install a messaging application.
* Does not anticipate changing address in the next 6 months.
* Understands spoken and written spanish language.
* Accepts to participate and signs the informed consent.

Exclusion Criteria:

* Communicative barriers.
* Addiction to other substances.
* Participation in another cessation program or other clinical trial during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Continuous tobacco abstinence at six months biochemically validated | Six months
  Patient declares to have smoked less than five cigarettes in the last six months and have less than 10 parts per million (ppm) of carbon monoxide in exhaled air measured by a Pico+TM Smokerlyzer® cooximeter

SECONDARY OUTCOMES:
Continuous tobacco abstinence at six months referred by patient | Six months
  Patient declares to have smoked less than five cigarettes in the last six months
Descriptive improvement in patient´s quality of life | Six months
  EuroQol 5D-5L questionary score descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Patient is asked to indicate health state by ticking the box next to the most appropriate statement in each dimension. This results in a 1-digit number that expresses the level selected for that dimension. Digits can be combined into a 5-digit number that describes the patient's health state.
Sujective improvement in patient´s quality of life | Six months
  EuroQol 5D-5L questionary score visual analogue scale (EQ VAS).
  EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. Can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
QALYs | Six months
  Quality-adjusted life years
Number of therapeutic contacts | Six months
  Number of contacts (therapist-patient or bot-patient) during the therapeutic process
Time spent in therapy | Six months
  Total amount of time spent (in minutes) during the therapeutic process

CONTACTS AND LOCATIONS:
Overall Officials: José F Ávila-Tomás, Doctor, Study Chair — GAP Madrid; Francisco J Ayesta-Ayesta, Doctor, Study Chair — Cantabria University; Francisco J Martínez-Suverbiola, Doctor, Study Chair — GAP Madrid
Locations (1):
- Eduardo Olano-Espinosa, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
No Plan has been developed

REFERENCES:
- [Derived] Olano-Espinosa E, Avila-Tomas JF, Minue-Lorenzo C, Matilla-Pardo B, Serrano Serrano ME, Martinez-Suberviola FJ, Gil-Conesa M, Del Cura-Gonzalez I; Dejal@ Group. Effectiveness of a Conversational Chatbot (Dejal@bot) for the Adult Population to Quit Smoking: Pragmatic, Multicenter, Controlled, Randomized Clinical Trial in Primary Care. JMIR Mhealth Uhealth. 2022 Jun 27;10(6):e34273. doi: 10.2196/34273. PMID 35759328
- [Derived] Avila-Tomas JF, Olano-Espinosa E, Minue-Lorenzo C, Martinez-Suberbiola FJ, Matilla-Pardo B, Serrano-Serrano ME, Escortell-Mayor E; Group Dej@lo. Effectiveness of a chat-bot for the adult population to quit smoking: protocol of a pragmatic clinical trial in primary care (Dejal@). BMC Med Inform Decis Mak. 2019 Dec 3;19(1):249. doi: 10.1186/s12911-019-0972-z. PMID 31796061